CLINICAL TRIAL: NCT01891838
Title: Transsphenoidal Surgery for Pituitary Adenomas: Influence of the Ventilation Mode on Intraoperative Bleeding
Brief Title: Mode of Ventilation and Bleeding During Transsphenoidal Surgery
Acronym: Vent-Hyp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/15; 2012-A00397-36 (Other: ANSM)
Record Dates: First submitted 2013-06-29; First posted 2013-07-03 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Surgery
Keywords: surgery; transsphenoidal surgery; pituitary adenoma; mechanical ventilation; bleeding
MeSH Terms: conditions — Pituitary Neoplasms; Hemorrhage

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volume controlled ventilation (Active Comparator): Volume controlled ventilation: tidal volume of 7 mL/kg ideal body weight, frequency of 12 cycles/minute, I/E ratio of 1:2, no positive end expiratory pressure. Ventilatory frequency is changed if necessary to maintain end-expiratory pressure of CO2 between 35 and 40 mmHg.
  Interventions: Procedure: Volume controlled ventilation
- Pressure-controlled ventilation (Experimental): initial pressure of 15 cm H2O, frequency of 12 cycles/minute, I/E ratio of 1:2, no positive end expiratory pressure. Pressure is modified to maintain a tidal volume of 7 mL/kg of ideal body weight and frequency ventilation is modified to maintain end-expiratory pressure of CO2 between 35 and 40 mmHg
  Interventions: Procedure: Pressure-controlled ventilation

INTERVENTIONS:
Procedure: Volume controlled ventilation
  Arms: Volume controlled ventilation
Procedure: Pressure-controlled ventilation
  Arms: Pressure-controlled ventilation

SUMMARY:
The risk of bleeding is important during transsphenoidal surgery. This study aims to find if the ventilation mode, controlled pressure and controlled volume, modifies the risk of bleeding.

DETAILED DESCRIPTION:
The risk of bleeding is important during transsphenoidal surgery. This study aims to find if the ventilation mode, controlled pressure and controlled volume, modifies the risk of bleeding.

* group Volume controlled ventilation: tidal volume of 7 mL/kg ideal body weight, frequency of 12 cycles/minute, I/E ratio of 1:2, no positive end expiratory pressure. Ventilatory frequency is changed if necessary to maintain end-expiratory pressure of CO2 between 35 and 40 mmHg.
* group Pressure-controlled ventilation: initial pressure of 15 cm H2O, frequency of 12 cycles/minute, I/E ratio of 1:2, no positive end expiratory pressure. Pressure is modified to maintain a tidal volume of 7 mL/kg of ideal body weight and frequency ventilation is modified to maintain end-expiratory pressure of CO2 between 35 and 40 mmHg.
* In both groups, the fraction of inspired oxygen is 50%. A recruitment maneuver is performed if the blood oxygen saturation became less than 92%.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Patients scheduled for transsphenoidal surgery for pituitary adenomas

Exclusion Criteria:

* Pregnancy
* Obesity (BMI> 35)
* Known respiratory disease
* Redo surgery
* Preoperative problem with hemostasis (antiplatelet or anticoagulant treatment; constitutional disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
intraoperative bleeding | 1 hour postoperatively
  intraoperative bleeding is estimated by the operator (always the same) as minimal (1), low (3), with no significant change in the conduct of the surgical procedure (5) with significant change in the conduct of surgical procedure (7). Intermediate levels are used to rate the levels of intermediate severity.

SECONDARY OUTCOMES:
generated plateau pressures | one hour after surgery
  mean ventilatory plateau pressure during surgery
realisation of predefined objectives of minute ventilation | one hour after surgery
  time spent with the predefined objectives of minute ventilation
changes of ventilation mode | one hour after surgery
  number of changes of ventilation mode
arterial desaturation | one hour after surgery
  number of episodes of arterial desaturation (SpO2 <92%) and lower arterial saturation during surgery
recruitment maneuver | one hour after surgery
  number of recruitment maneuver
duration of the surgical procedure | one hour after surgery
  duration from surgical incision to end of the surgical procedure
endocrine healing | three months after surgery
  return to a low level of the abnormal endocrin abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hôpital Foch
Locations (1):
- Hopital Foch, Suresnes, France

REFERENCES:
- [Derived] Le Guen M, Paternot A, Declerck A, Feliot E, Gayat E, Gaillard S, Fischler M. Impact of the modality of mechanical ventilation on bleeding during pituitary surgery: A single blinded randomized trial. Medicine (Baltimore). 2019 Sep;98(38):e17254. doi: 10.1097/MD.0000000000017254. PMID 31567997